CLINICAL TRIAL: NCT05390788
Title: Effect of Neuromuscular Bands on Knee Joint Position Sense in Healthy Subjects
Brief Title: KinesioTaping on Knee Joint Position Sense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Saude do Alcoitao (Other)
Responsible Party: Principal Investigator, João Afonso Correia, Principal Investigator, Afonso Correia, Escola Superior de Saude do Alcoitao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 07/2022
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: Proprioception; Joint Position Sense; Neuromuscular Bands; Isokinetic Dynamometer; Kinesiotaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Joint Position Sense is measured in 6 different moments. 1st Moment: Measurement with no intervention; 2nd Moment: 5 days later, imediately before intervention (kinesiotaping/neuromuscular bands); 3rd Moment: Imediately after intervention; 4th Moment: 5 days after the previous measurement, with kinesiotape still applied; 5th Moment: Measurement imediately after removing kinesiotape; 6th Moment: 5 days after the previous measurement, with no intervention (follow-up)
  Interventions: Other: Application Of Neuromuscular Bands; Kinesio Taping
- Control Group (No Intervention): 4 Measurements with no intervention, with a 5 day interval between

INTERVENTIONS:
Other: Application Of Neuromuscular Bands; Kinesio Taping — Kinesio tape is a specialized elastic and adherent adhesive tape that mimics the elasticity of skeletal muscle, in that it can be extended up to 140% of its original length, before application to the skin, without allowing restrictions in the range of motion. of structures. Subsequently, it provides a tensile (shear) force on the skin, consisting of a fabric with special characteristics, such as air permeability and water resistance, and can be used for repeated days. Kinesio will be applied from a point 10 cm below the anterior superior iliac spine and divided in a "Y" shape above the patella, ending at the tibial tuberosity; from the upper third of the medial thigh to the medial border of the patella; from the greater trochanter of the femur, ending at the lateral margin of the patella.
  Other Names: Kinesiotaping
  Arms: Experimental Group

SUMMARY:
The aim of this study is to evaluate the effect of kinesio tape (Neuromuscular bands) application on knee joint position sense. The investigators intend to evaluate, trough the use of an isokinetic dynamometer, the sensation of active and passive joint position sense of the knee joint, before, during and after the application of kinesio tape in different periods, and to verify if there is any noticeable change. The guiding question is presented as the following: "Does the application of kinesio tape influence the knee joint position sense in healthy young adults?".

The hypothesis of this study is represented as follows:

H1: Kinesio tape application improves knee joint position sensation in healthy young adults.

H0: Kinesio tape application has no influence on knee joint sensation and position in healthy young adults.

DETAILED DESCRIPTION:
As mentioned before, the aim of this study is to evaluate the effect of kinesio tape (Neuromuscular bands) application on knee joint position sense. After explaining the objectives and procedures of the study, the subjects will sign an informed consent. Afterwards, the sample subjects will be randomly divided into two groups, the experimental group and the control group. Joint position sense will be measured at four different times in the control group and at 6 different times in the experimental group. In the first moment of data collection, anthropometric data of the participants will be measured, namely weight and height, and a sociodemographic questionnaire will be completed. Then, the identification of the dominant side of the individual will be carried out, through the step test, in which we ask the individual to climb a step 3 times and through the ball kick test. All subjects will always have to carry out measurements in shorts and t-shirts, completely barefoot. The intervention, in the experimental group, will consist of the application of neuromuscular bands on the dominant lower limb. No intervention will be performed in the control group. A physical therapist will be in charge of applying the neuromuscular bands to the participants and another physical therapist will take measurements of joint position sense.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals from 18 to 35 years old

Exclusion Criteria:

* Musculoskeletal condition in the dominant lower limb 3 months before the beggining of the study;
* Central and Periferical Nervous System alteration;~
* Pain In the dominant lower limb;
* History of fracture on the dominant lower limb;
* Adverse reactions to ahesive materials;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Joint Position Sense | 30 minutes
  The difference of error in degrees was calculated to show changes in error from the target angles over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde do Alcoitão, Cascais, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No